CLINICAL TRIAL: NCT01728129
Title: Comparison of the Defense Automated Neurobehavioral Assessment (DANA) Tool to the Military Acute Concussion Evaluation (MACE) in the Evaluation of Suspected Acute Concussion
Brief Title: DANA Compared to MACE in Evaluation of Suspected Acute Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, jack tsao, Director, TBI Programs, United States Department of Defense
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: M-10228
Record Dates: First submitted 2012-11-08; First posted 2012-11-16 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Brain Concussion; Traumatic Brain Injury
Keywords: Concussion; Mild traumatic brain injury; DANA; MACE
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic | interventions — omega-Chloroacetophenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concussed (Experimental): Subjects who are diagnosed with a concussion by a clinician will be assessed with the MACE and DANA Rapid every 24 hours for up to 72 hours post-injury.
  Interventions: Device: DANA Rapid; Other: MACE
- Non-concussed (Active Comparator): Subjects will have been exposed to a potentially concussive event but be clinically evaluated and found not to have sustained a concussion. Control subjects from this arm will take both the MACE and DANA Rapid twice: once within 24 hours of potentially concussive event, and again on the day of return to duty.
  Interventions: Device: DANA Rapid; Other: MACE

INTERVENTIONS:
Device: DANA Rapid — The DANA Rapid is a neurocognitive test self-administered on a small handheld computer. The DANA Rapid subtests measure simple reaction time, procedural reaction time, and reaction time sensitivity.
Other: MACE — The MACE is currently the only standardized and Department of Defense-designated method for the initial evaluation of suspected concussion in military operational settings. The MACE documents the history of the injury-causing incident; assesses cognitive deficits in orientation, immediate memory, concentration, and delayed recalls; and involves a neurological screening by a clinician.

SUMMARY:
The purpose of this study is to compare the sensitivity of the DANA Rapid exam with the MACE cognitive score. The primary hypothesis is that the DANA Rapid exam will be more sensitive for detecting impaired cognitive performance than the MACE cognitive score in the setting of a clinical diagnosis of concussion at the point of injury in the combat setting. A secondary purpose of this study is to examine a serial performance on the DANA Rapid exam in those subjects diagnosed with a concussion. The secondary hypothesis is that the DANA Rapid exam will show improvements in performance during the recovery period after concussion.

DETAILED DESCRIPTION:
In Operations Iraqi Freedom and Enduring Freedom (OIF/OEF), over 60% of combat casualties have been the result of explosive blasts, and many of these critical injuries involve trauma to the head. As a result, traumatic brain injury (TBI) has been deemed a "signature wound" of OIF and OEF. The symptoms of head injuries, particularly of concussion/mild TBI (mTBI), can be sever but subtle, suggesting that early and accurate diagnosis is paramount to a wounded warrior's appropriate medical care. Most first providers in the war theater are medics who could benefit from an improved diagnostic test to better identify service members with concussion/mTBI. The MACE cognitive test is heavily weighted towards memory, is not 100% specific, and does not preclude a diagnosis of concussion being rendered despite a score in the normal range. Thus, an objective test of neurocognitive function, such as the DANA Rapid, that can be rapidly administered in theater by a combat medic would be highly beneficial to accurate clinical diagnosis and timely treatment. The results of the present study will provide information on the predictive value of the newly developed DANA handheld computer in assisting in the diagnosis of concussion in service members who have been blast exposed. If the DANA Rapid exam proves to be equally or more accurate than the MACE in detecting cognitive deficits, these tests and the handheld computer will also contribute to improved health care for service members by minimizing the time between injury and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military personnel
* Glasgow Coma Scale (GCS)score of 15, as assessed by the study member at the time of clinical evaluation following involvement in a mandatory event.
* Willingness to participate in the study, ability to communicate and comply with the study protocol and ability to provide informed consent

Exclusion Criteria:

* GCS score of less than 15

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 72 hours from initial injury
  The primary hypothesis is that an abnormal score on the DANA Rapid will positively identify a greater proportion of concussed individuals than an abnormal cognitive score on the MACE would. Conversely, scores within normal range on the DANA Rapid should be able to rule out cognitive deficits more accurately than a normal score on the MACE

SECONDARY OUTCOMES:
Serial Performance | 72 hours from initial injury
  The secondary hypothesis of the study is that scores on the DANA Rapid exam will improve over time as the subject recovers from concussion.

CONTACTS AND LOCATIONS:
Overall Officials: Jack W. Tsao, MD, DPhil, Principal Investigator — U.S. Navy Bureau of Medicine and Surgery (BUMED)
Locations (1):
- Concussion Restoration Care Center, Camp Leatherneck, Afghanistan